CLINICAL TRIAL: NCT00172692
Title: Observation and Evaluation of Chewing Velocity Changes on Soft Food Chewing Efficiency
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9361701237
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2006-12-15 (Estimated); Status verified 2005-06

CONDITIONS: Healthy; Mastication
Keywords: Chewing efficiency,; Gum chewing; Chewing velocity; Occlusal surface area; EMG; Jaw movement

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
Soft food chewing does not require strong bite force. The number of chewing strokes and occlusal surface area of the posterior teeth are more important. Clinically, reduction of occlusal surface to protect the abutments of a fixed or removable partial denture or the implant supported teeth is often necessary. If a certain chewing ability is maintained with reduced occlusal area, changing chewing velocity might help. For this hypothesis, the effect of chewing velocity on soft food chewing ability would be observed first. The purpose of this study is to evaluate the deliberately changed chewing gum chewing velocity on the chewing ability of healthy subjects whose dental occlusal surface area is known. Twenty dental students (10 men and 10 women with an age range of 20-30 years) with healthy masticatory systems and complete dentition will be asked to chew HA containing chewing gum with habitual side teeth at the cycle time of 0.5 sec, 1.0 sec and 1.5 sec for 30, 40, and 50 times. Jaw movement, tooth contact, and muscle activities will be observed during chewing gum chewing. The distribution of HA particles in the gum bolus after each chewing session will be measured and regarded as the chewing efficiency of that subject. Occlusal surface area of the maxillary posterior teeth, chewing rate, chewing time, muscle activity and jaw lateral displacement will be related to the chewing efficiency with multiple regression analysis. The effects of practice due to changing of chewing rate will also be evaluated.

DETAILED DESCRIPTION:
1. HA containing chewing gum with habitual side teeth at the cycle time
2. The distribution of HA particles in the gum bolus after each chewing session will be measured and regarded as the chewing efficiency of that subject.

National Taiwan University Hospital, National Science Council

ELIGIBILITY:
Inclusion Criteria:

* Dental students
* Healthy masticatory system

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Start 2004-07; Study Completion 2004-08

CONTACTS AND LOCATIONS:
Overall Officials: Yuh-Yuan Shiau, Professor, Study Chair — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan